CLINICAL TRIAL: NCT07319884
Title: The Role of Fluoride Varnish Application in Preventing White Spot Lesions During Clear Aligner Treatment: A Controlled Split-Mouth Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Jalal Alshami, Dentist Jalal-Alshami, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Mansoura-university
Record Dates: First submitted 2025-12-20; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: White Spot Lesion

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- White spot lesion with fluoride varnish application during clear Aligner therapy (Experimental): Intervention Group (Test Side):
  • Application of a preventive fluoride varnish on the indicated side of the mouth before clear aligner fitting.
  Interventions: Other: White spot lesion with fluoride varnish application
- White spot lesion without fluoride varnish application during clear Aligner therapy (Active Comparator): Control Group (Control Side): No application of fluoride varnish.
  Interventions: Other: White spot lesion without fluoride varnish application

INTERVENTIONS:
Other: White spot lesion with fluoride varnish application — Application of fluoride varnish at the cervical third of labial surface or around the attachment if present
  Arms: White spot lesion with fluoride varnish application during clear Aligner therapy
Other: White spot lesion without fluoride varnish application — No fluoride varnish application at the cervical third of the labial surface or around the attachment if present
  Arms: White spot lesion without fluoride varnish application during clear Aligner therapy

SUMMARY:
aim of study: is to compare the effect of the fluoride varnish application on the prevention of white spot lesions (WSLs) during clear aligner therapy

Design Details: Each participant will have one side of the mouth assigned to the fluoride varnish intervention, while the contralateral side will serve as the control without fluoride varnish.

Outcomes:

Primary outcome: Incidence and Severity of White Spot Lesions Measured before and after six months using Laser fluorescence (DIAGNOdent)

Secondary Outcome:

Periodontal Ligament (PDL) Health using pocket Depth Index (PDI) Gingival Bleeding and Inflammation using bleeding on Probing Index (BOP)

DETAILED DESCRIPTION:
aim of study: is to compare the effect of the fluoride varnish application on the prevention of white spot lesions (WSLs) during clear aligner therapy in comparison to a split mouth-controlled group

Sample size calculation:

The sample size was calculated using G* power software (version3.1.9.7) and was designed to have a power of 85% assuming a type I statistical error of 5% and a one tailed statistical test with an effect size f= 0.7730012 based on the study of Najafi et al. The means and standard deviation of the DIAGNOdent score of the varnish and control groups after six months were 1.23 ±0.45 and 1.78±0.90. The calculated sample size will be 25 patients. The sample size will be increased to include 30 patients to avoid any drop out.

Material and methods:

1. Initial Oral Scan:

   • A 3D oral scan of the arch to be treated will be performed using a digital intraoral scanner
2. Aligner Fabrication:

   * aligners will be fabricated using thermoforming techniques.
   * A clear aligner sheet (e.g.Duran) is heated and vacuum or pressure-formed over the 3D-printed model, then trimming followed by finishing and polishing
3. Interventions

Intervention Group (Test Side):

• Application of a preventive fluoride varnish (Charm varnish) on the indicated side of the mouth before clear aligner fitting.

Control Group (Control Side):

* Without application of fluoride varnish 4. Aligner Placement:
* The aligners will be fitted, and patients will wear them continuously, except during eating and brushing.

Outcome Measures:

Primary Outcome:

• Incidence and Severity of White Spot Lesions Measured before and after six months using Laser fluorescence (DIAGNOdent)

Secondary Outcome:

1. Periodontal Ligament (PDL) Health using:

   * Pocket Depth Index (PDI)
2. Gingival Bleeding and Inflammation using:

   * Bleeding on Probing Index (BOP)

Randomization and Application Site

To minimize bias, the side of the maxillary arch (right or left upper side) for fluoride varnish application was randomly assigned for each of the patients using a computer-generated randomization sequence

Inclusion and Exclusion Criteria Eligible participants were patients aged 16-24 years, representing the typical demographic for clear aligner therapy and ensuring biological consistency in terms of tooth development and orthodontic response. All participants were required to be in good general and oral health to minimize confounding factors related to systemic or oral disease, to present with mild dental crowding in each arch to standardize treatment complexity, and to have full eruption of all permanent teeth excluding third molars to allow consistent varnish application and assessment. Patients were excluded if they had a known allergy or hypersensitivity to fluoride-containing materials, systemic conditions that could affect tooth movement (such as diabetes or bone metabolism disorders), cleft lip and/or palate or other craniofacial anomalies, a history of previous orthodontic treatment, or clinical evidence of dental fluorosis, as these factors could alter enamel characteristics, orthodontic response, or lesion assessment and thereby introduce bias into the study outcomes.

Duration of the study:

• This study is suggested to be finished in 18 months

ELIGIBILITY:
Inclusion Criteria:

* patients aged 16-24 years.
* Good general and oral health.
* Mild dental crowding per arch (≤ 4 mm).
* Eruption of all permanent dention excluding third molar

Exclusion Criteria:

* Allergy to fluoride material
* Systemic conditions affecting tooth movement (e.g., diabetes, bone disorders).
* Patients with Cleft lip and palate
* Previous orthodontic treatment
* dental fluorosis.
* hypocalcified teeth or visible demineralization

Ages: 16 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 25 (Actual)
Dates: Start 2025-06-25 (Actual); Primary Completion 2027-01-25 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Incidence and Severity of White Spot Lesions | Six months
  Incidence and Severity of White Spot Lesions Measured before and after six months using Laser fluorescence (DIAGNOdent)

SECONDARY OUTCOMES:
Periodontal Ligament (PDL) Health | Six moths
  Health using pocket Depth Index (PDI)
Gingival Bleeding and Inflammation | Six months
  using bleeding on Probing Index (BOP)

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of dentistry Mansoura University, Al Mansurah, Egypt